CLINICAL TRIAL: NCT07073365
Title: A Prospective Cohort Observational Study of Local Therapy for the Primary Tumor in EGFR-Mutant Advanced Non-Small Cell Lung Cancer Following Osimertinib Plus Chemotherapy (FLAURA2 Regimen)
Brief Title: Bolstering Outcomes After Induction With Osimertinib Plus Chemotherapy Through Optimized Site-Directed Primary Tumor Therapy (BOOST Trial)
Acronym: BOOST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNU-002
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer; Epidermal Growth Factor Receptor
Keywords: Non-Small Cell Lung Cancer; EGFR Mutation; FLAURA2; Osimertinib; Local Therapy; Surgery; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Single-arm study with local therapy after systemic treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Local Therapy Arm (Experimental): Patients with EGFR-mutant advanced non-small cell lung cancer who achieve disease control after first-line osimertinib plus chemotherapy (FLAURA2 regimen) will receive local therapy (surgery or radiotherapy) to the primary tumor. The study will evaluate clinical outcomes including progression-free survival, overall survival, and treatment-related toxicity.
  Interventions: Other: Local Therapy (Surgery or Radiotherapy)

INTERVENTIONS:
Other: Local Therapy (Surgery or Radiotherapy) — Patients will receive local therapy, either surgical resection or radiotherapy, to the primary lung tumor following disease control after first-line treatment with osimertinib plus platinum-based chemotherapy (FLAURA2 regimen). The specific modality (surgery or radiotherapy) will be determined based on tumor characteristics, patient condition, and multidisciplinary team assessment.

SUMMARY:
This is a single-arm, open-label, phase II study evaluating the clinical outcomes of local therapy (surgery or radiotherapy) to the primary tumor in patients with EGFR-mutant advanced non-small cell lung cancer (NSCLC) who have achieved disease control following first-line treatment with the FLAURA2 regimen (osimertinib plus platinum-based chemotherapy). The primary objective is to assess the median progression-free survival (PFS) after local therapy.

DETAILED DESCRIPTION:
This prospective, single-arm, multicenter observational study is designed to estimate the median progression-free survival (PFS) in patients with EGFR-mutant advanced non-small cell lung cancer (NSCLC) who receive salvage local treatment after achieving disease control with first-line osimertinib plus chemotherapy. A total of 70 patients will be enrolled. The primary endpoint is median PFS, and the sample size was calculated to ensure that the 95% confidence interval around the estimated median has a width of no more than ±3 months, using Greenwood's approximation. Patients will be followed for a minimum of 24 months after the last enrollment, with an overall study duration of up to 72 months.

ELIGIBILITY:
<Inclusion Criteria>

Participants must meet all of the following criteria to be eligible:

1. Age ≥ 20 years at the time of consent.
2. Histologically or cytologically confirmed diagnosis of non-small cell lung cancer (NSCLC).
3. Presence of activating EGFR mutation (exon 19 deletion or L858R).
4. Stage IV (metastatic) NSCLC at initial diagnosis.
5. Completion of four cycles of first-line osimertinib plus platinum-based chemotherapy (FLAURA2 regimen).
6. Radiologic evidence of disease control (complete response, partial response, or stable disease) after systemic therapy.
7. Residual primary lung tumor suitable for local therapy (surgery or radiotherapy), as determined by multidisciplinary evaluation.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Adequate organ function based on institutional laboratory criteria.
10. Ability to understand and willingness to provide written informed consent.

<Exclusion Criteria>

Participants will be excluded if they meet any of the following criteria:

1. Radiologic or clinical evidence of progressive disease during first-line osimertinib-chemotherapy.
2. Extensive, unresectable metastatic disease not amenable to local therapy.
3. Untreated or clinically unstable brain metastases.
4. Known contraindications to surgery or radiotherapy.
5. Active second malignancy requiring concurrent treatment.
6. Any condition that, in the opinion of the investigator, would interfere with study participation or interpretation of results.
7. Pregnancy or breastfeeding at the time of enrollment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival (PFS) | Up to 60 months (through June 30, 2030; patients followed for ≥24 months after last enrollment)
  Time from the initiation of local therapy to the date of radiographic or clinical disease progression or death from any cause, whichever occurs first. Median PFS will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 72 months (through June 30, 2031)
  Time from initiation of local therapy to death from any cause. OS will be estimated using the Kaplan-Meier method, and survival rates at predefined time points (e.g., 2-year OS) will also be reported.
Local Control Rate | Up to 60 months (through June 30, 2030)
  Proportion of patients without local tumor progression at the treated site(s), assessed radiographically. Local control will be evaluated, including the 24-month local control rate.
Adverse events (AEs) | Up to 60 months (through June 30, 2030)
  Incidence, type, and severity of treatment-related adverse events will be recorded. Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Hyun Kim, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Kim MH, Seong H, Kim SH, Eom JS. Local consolidative therapy for the primary tumor in EGFR-mutant advanced non-small cell lung cancer following osimertinib plus chemotherapy: a protocol for a single-arm, open-label, phase 2 trial. Transl Lung Cancer Res. 2025 Oct 31;14(10):4666-4674. doi: 10.21037/tlcr-2025-922. Epub 2025 Oct 29. PMID 41234591